CLINICAL TRIAL: NCT04186351
Title: Efficacy of Providing an Automated Notification Service, the "Encounter Notification Service" Via the eHRSS for Home-based Care and Services Provided by Community Healthcare Providers for the Elderly: A 12-month Randomized Controlled Trial
Brief Title: Electronic Health Record Sharing System (eHRSS) Encounter Notification Service Pilot Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Calvin Or, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MYCARER 20191108
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Home-dwelling Elderly; Health Care Recipient
Keywords: automated notification service; community healthcare providers; randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encounter notification service (Experimental): For participants randomized to the intervention group, their encounter information stored in the eHRSS will be provided to the SCHSA via the automated notification service. Healthcare professionals of the SCHSA would access the electronic health record and provide caring support and services via telephone calls during the 12-month study period.
  Interventions: Behavioral: Encounter notification service
- Usual care service (No Intervention): For participants randomized in the control group, no notification will be sent to the SCHSA. Usual care service will be provided during the 12-month study period. In addition, each control participant will receive placebo phone calls at least once every three months (e.g., the calls could be about greeting and general checking).

INTERVENTIONS:
Behavioral: Encounter notification service — The caring support and services provided by SCHSA will consist of multiple components, including standard call & care center support, medical appointment reminder, assistance to reschedule appointment, follow-up calls with either nurse or health workers to monitor health situation of service recipients, assessing needs of service recipient for elderly home care and/or rehabilitation services, providing elderly home care and/or rehabilitation services based on assessment, assessing needs of service recipient for emotional and community support, providing additional emotional support via either social calls by volunteers or counseling by social workers, and making referrals for community support services.
  Arms: Encounter notification service

SUMMARY:
This study evaluates the value of the automated notification service that allows more timely information access and sharing. A 12-month RCT will be conducted to determine the efficacy of the provision of the service to an elderly care and service provider in improving care and health outcomes of the elderly. Researchers will also examine whether the notification service will better support the carers for the coordination and prioritization of care and service delivery.

DETAILED DESCRIPTION:
A research team at the University of Hong Kong is commissioned to conduct a study of the efficacy of providing an automated notification service, i.e., the "Encounter Notification Service," via the Electronic Health Record Sharing System (eHRSS) to an elderly caring and service provider that aims to facilitate more timely provision and coordination of healthcare services for home-dwelling elderly. With the access to the automated notification service containing up-to-date encounter information of the elderly in the eHRSS (e.g. discharge date from the public hospital, outpatient appointments), it is expected that the elderly caring and service provider can improve its allocation of resources and prioritize the provision of service to elderly patients who are in need, i.e., during the transition of care. As a result, the caring support and services provided by the elderly caring and service provider to the elderly can be more timely and effective, and an improvement in patient health outcomes can be expected.

To obtain evidence to determine the value of the automated notification service, a systematic study of the efficacy is suggested. Thus, researchers set out to conduct a 12-month randomized controlled trial (RCT) to examine whether the provision of the automated notification service to the caring and service provider will result in improvements in care and health outcomes of the elderly. Also, researchers will assess whether the notification service will better support the carers for the coordination and prioritization of care and service provision and improve workflow and administrative procedures amongst different sectors.

In this pilot study, the Senior Citizen Home Safety Association (SCHSA) is the participated elderly caring and service provider.

ELIGIBILITY:
Inclusion Criteria:

* are aged 18 years or older
* have registered in eHRSS as healthcare recipients and given consent for sharing their records in the eHRSS with the SCHSA
* are able to understand spoken Cantonese

Exclusion Criteria:

* with mental incapacity
* with hearing difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-12-14 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in the number of Accident and Emergency (A&E) visits | from baseline to 6 and 12 months

SECONDARY OUTCOMES:
changes in the number of non-attendance to outpatient appointments | from baseline to 6 and 12 months
changes in the number of unplanned hospitalizations | from baseline to 6 and 12 months
changes in the number of 30-day unplanned readmissions | from baseline to 6 and 12 months
changes in the stability of health condition | from baseline to 6 and 12 months
  measured by a questionnaire with items on a 5-point Likert scale ranging from 1 (worse outcome) to 5 (better outcome)
changes in the understanding of the arrangement of outpatient appointments | from baseline to 6 and 12 months
  measured by a questionnaire with items on a 5-point Likert scale ranging from 1 (worse outcome) to 5 (better outcome)
changes in the elderly's perceptions of the services | from baseline to 6 and 12 months
  measured by a questionnaire with items on a 5-point Likert scale ranging from 1 (worse outcome) to 5 (better outcome)

OTHER OUTCOMES:
changes in the carers' perceptions of the impacts of the notification service | from baseline to 6 and 12 months
  A questionnaire survey will be conducted to assess carers' perceptions of the automated notification service on care coordination and prioritization, workflow, and administrative procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Kalun Or, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Senior Citizen Home Safety Association, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sommers LS, Marton KI, Barbaccia JC, Randolph J. Physician, nurse, and social worker collaboration in primary care for chronically ill seniors. Arch Intern Med. 2000 Jun 26;160(12):1825-33. doi: 10.1001/archinte.160.12.1825. PMID 10871977
- [Background] Mizrahi T, Abramson JS. Collaboration between social workers and physicians: perspectives on a shared case. Soc Work Health Care. 2000;31(3):1-24. doi: 10.1300/J010v31n03_01. PMID 11101162
- [Background] Beck A, Scott J, Williams P, Robertson B, Jackson D, Gade G, Cowan P. A randomized trial of group outpatient visits for chronically ill older HMO members: the Cooperative Health Care Clinic. J Am Geriatr Soc. 1997 May;45(5):543-9. doi: 10.1111/j.1532-5415.1997.tb03085.x. PMID 9158573
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163